CLINICAL TRIAL: NCT06859424
Title: A Platform Protocol to Investigate Post-Transplant Cyclophosphamide-Based Graft-Versus-Host Disease Prophylaxis in Patients With Hematologic Malignancies Undergoing Mismatched Unrelated Donor Peripheral Blood Stem Cell Transplantation
Acronym: ACCELERATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCELERATE
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: AML (Acute Myelogenous Leukemia); Acute Lymphoid Leukemia (ALL); Acute Leukemia (Category); MDS (Myelodysplastic Syndrome); CML (Chronic Myelogenous Leukemia); CLL (Chronic Lymphocytic Leukemia); Prolymphocyctic Leukemia; Chronic Myelomonocytic Leukemia (CMML); Myeloproliferative Neoplasm (MPN); Lymphoma; Myelofibrosis
Keywords: ACCELERATE; ACCEL-001; ACCEL-002
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, B-Cell; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Lymphoma; Primary Myelofibrosis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: A randomized, multi-center, prospective, controlled platform trial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control/SOC (Experimental): Shared comparator control group
  Interventions: Drug: Conditioning Regimen A; Drug: Conditioning Regimen B; Drug: Conditioning Regimen C; Drug: Conditioning Regimen D; Drug: Conditioning Regimen E; Procedure: Hematopoietic Cell Transplantation; Drug: PTCy (50 mg/kg D3, D4); Drug: Post-transplant Tacrolimus; Drug: Post-transplant Mycophenolate mofetil; Drug: Supportive Care: Growth Factors; Procedure: Supportive Care: Blood Products; Other: Supportive Care: Infection Prophylaxis; Other: Supportive Care: Intravenous immune globulin (IVIG); Drug: Supportive Care: Seizure prophylaxis; Other: Supportive Care: Monitoring and management of CRS; Other: Study treatment compliance; Other: Prohibited Concomitant Therapy; Other: Permitted Concomitant Therapy
- ACCEL-001 (Experimental): Intervention 1
  Interventions: Drug: Conditioning Regimen A; Drug: Conditioning Regimen B; Drug: Conditioning Regimen C; Drug: Conditioning Regimen D; Drug: Conditioning Regimen E; Procedure: Hematopoietic Cell Transplantation; Drug: PTCy (25 mg/kg D3, D4); Drug: Post-transplant Tacrolimus; Drug: Post-transplant Abatacept; Drug: Supportive Care: Growth Factors; Procedure: Supportive Care: Blood Products; Other: Supportive Care: Infection Prophylaxis; Other: Supportive Care: Intravenous immune globulin (IVIG); Drug: Supportive Care: Seizure prophylaxis; Other: Supportive Care: Monitoring and management of CRS; Other: Supportive Care: Prophylaxis against infections; Other: Study treatment compliance; Other: Prohibited Concomitant Therapy; Other: Permitted Concomitant Therapy
- ACCEL-002 (Experimental): Intervention 2
  Interventions: Drug: Conditioning Regimen A; Drug: Conditioning Regimen B; Drug: Conditioning Regimen C; Drug: Conditioning Regimen D; Drug: Conditioning Regimen E; Procedure: Hematopoietic Cell Transplantation; Drug: PTCy (25 mg/kg D3, D4); Drug: Post-transplant Tacrolimus; Drug: Post-transplant Mycophenolate mofetil; Drug: Post-transplant Ruxolitinib; Drug: Supportive Care: Growth Factors; Procedure: Supportive Care: Blood Products; Other: Supportive Care: Infection Prophylaxis; Other: Supportive Care: Intravenous immune globulin (IVIG); Drug: Supportive Care: Seizure prophylaxis; Other: Supportive Care: Monitoring and management of CRS; Drug: Supportive Care: Prophylaxis against infections; Other: Supportive Care: Lipid elevations; Other: Study treatment compliance; Other: Prohibited Concomitant Therapy; Other: Permitted Concomitant Therapy

INTERVENTIONS:
Drug: Conditioning Regimen A — Busulfan and fludarabine
  Recommended schedule as below:
  * Days -6 to -3: Busulfan ≥ 9 mg/kg total dose (IV or PO) with pharmacokinetic (PK) monitoring recommended as per institutional practice to achieve a daily area under the curve (AUC) target of 4800-5300 μM*min47 or busulfan plasma exposure units (BPEU) 19.7-21.75 mg x h/L48.
  * Days -6 to -2: Flu 30 mg/m2/day (adjusted for renal function) is administered over a 30-60 minute IV infusion (maximum cumulative dose, 150 mg/m2).
Drug: Conditioning Regimen B — Fludarabine and TBI The recommended fludarabine plus TBI regimen is the following:
  * Days -7, -6 and -5: Flu (30 mg/m2/day, maximum cumulative dose, 90 mg/m2), IV
  * Days -4 to -1: TBI (150 cGy administered twice daily, 1200 cGy total dose)
    * Radiation sources, dose rates, and shielding follow institutional practice.
    * Although not required, it is recommended that palifermin be used to mitigate the risk of mucosal toxicity with this regimen.
Drug: Conditioning Regimen C — Fludarabine and busulfan (Flu/Bu)
  The recommended Flu/Bu regimen is the following:
  * Days -6 to -2: Flu (30 mg/m2/day, recommended total dose of 150 mg/m2, but not exceeding 180 mg/m2), IV Busulfan options
  * Days -5 to -4: Busulfan without PK - Busulfan 3.2 mg/kg/day IV or oral equivalent; total dose of 6.4 mg/kg IV or oral equivalent respectively
  * Days -5 to -4: Busulfan with PK - target doses to AUC of 4000 μMol/min or BPEU of 16.43 mg x h/L (total BPEU of 65.72 mg x h/L) or less is allowed.
Drug: Conditioning Regimen D — Fludarabine and melphalan (Flu/Mel)
  The recommended Flu/Mel regimen is the following:
  * Days -7 to -3: Flu (30 mg/m2/day or 25 mg/m2/day, total dose of 125-150 mg/m2), IV
  * Day -1: Mel (100-140 mg/m2 IV for recipients aged 18-59; dose of melphalan cannot exceed 100mg/m2 if age 60 or older or calculated glomerular filtration rate (GFR) is <60 ml/min), IV
Drug: Conditioning Regimen E — Fludarabine/cyclophosphamide/total body irradiation (Flu/Cy/TBI)
  The recommended Flu/Cy/TBI regimen is the following:
  * Days -6 to -5: Cy (14.5 mg/kg/day IV, total dose of 29 mg/kg, or single dose 50 mg/kg on Day -6 [Minnesota regimen])
  * Days -6 to -2: Flu (30 mg/m2/day, total dose of 150 mg/m2) IV
  * Day -1: TBI 200 cGy single dose Hydration and Mesna may be administered per institutional standards. For recipients of RIC/NMA AND donors matched at <7/8, consider the addition of TBI 200-300cGy for the Flu/Bu and Flu/Mel regimens to mitigate the risk of primary graft failure.
Procedure: Hematopoietic Cell Transplantation — * On Day 0, the donor PBSC graft is infused.
  * Donor PBSC will be collected per NMDP/donor registry policies with a target viable CD34+ cell dose of at least 4 × 106 /kg recipient weight (actual, ideal, or adjusted ideal per institutional practice).
  * Dose of CD34+ cells/kg and CD3 cells/kg infused will be recorded.
  * If the donor PBSC graft is cryopreserved prior to the start of conditioning, follow institutional practices to ensure a sufficient cell dose is available for infusion after thawing.
  * The graft cannot be manipulated ex vivo to deplete T cells.
Drug: PTCy (50 mg/kg D3, D4) — Cyclophosphamide (50mg/kg ideal body weight (IBW); [if actual body weight (ABW) < IBW, use ABW]) will be given on Day +3 (between 60 and 72 hours after the start of the PBSC infusion) and on Day 4 post HCT (approximately 24 hours after Day +3 cyclophosphamide). Cyclophosphamide will be given as an intravenous (IV) infusion over 1-2 hours (depending on volume), or according to institutional standards. Hydration pre- and post- cyclophosphamide and Mesna administration will be given per institutional standards.
  No systemic immunosuppressive agents are given until at least 24 hours after the completion of the PTCy. This includes corticosteroids as anti-emetics but excludes any drugs listed in section 7.9.1.
  Azoles (e.g., posaconazole or voriconazole) must be delayed from beginning of conditioning through completion of Day 4 PTCy dose to avoid potential drug-drug interactions with cyclophosphamide that could lead to increased toxicity.
  Arms: Control/SOC
Drug: PTCy (25 mg/kg D3, D4) — Cyclophosphamide (25mg/kg ideal body weight (IBW); [if actual body weight (ABW) < IBW, use ABW]) will be given on Day +3 (between 60 and 72 hours after the start of the PBSC infusion) and on Day 4 post HCT (approximately 24 hours after Day +3 cyclophosphamide). Cyclophosphamide will be given as an intravenous (IV) infusion over 1-2 hours (depending on volume), or according to institutional standards. Hydration pre- and post- cyclophosphamide and Mesna administration will be given per institutional standards.
  No systemic immunosuppressive agents are given until at least 24 hours after the completion of the PTCy. This includes corticosteroids as anti-emetics but excludes any drugs listed in Table 4 and Table 5 in Section 7.1.
  Azoles (e.g., posaconazole or voriconazole) must be delayed from beginning of conditioning through completion of Day 4 PTCy dose to avoid potential drug-drug interactions with cyclophosphamide that could lead to increased toxicity.
  Arms: ACCEL-001; ACCEL-002
Drug: Post-transplant Tacrolimus — Tacrolimus will be given per institutional practices, at a dose of 0.05 mg/kg per os (PO) or an IV dose of 0.03 mg/kg of IBW starting on Day + 5. The dose of tacrolimus may be rounded to the nearest 0.5 mg for oral formulations. Subsequent dosing will be based on blood levels per institutional guidelines with a suggested range of 5-12 ng/mL. If subjects are on medications which alter the metabolism of tacrolimus (e.g., concurrent CYP3A4 inhibitors), the initial starting dose and subsequent doses should be altered as per institutional practices. Tacrolimus taper is recommended to be initiated at 100 days post HCT if there is no evidence of active GVHD and ended by Day + 180 post HCT.
Drug: Post-transplant Mycophenolate mofetil — MMF will be given at a dose of 15 mg/kg 3 times daily (TID) (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1g TID, IV or PO). MMF prophylaxis will start Day + 5 and continue until Day + 35 post-transplant, at which time it should be discontinued (no taper necessary). Study site investigators may modify dose/taper early if clinically indicated for the study subject. Dose rounding may be done per institutional practice.
  Arms: ACCEL-002; Control/SOC
Drug: Post-transplant Abatacept — Abatacept will be given at a dose of 10 mg/kg with a maximum of 1000 mg.
  Arms: ACCEL-001
Drug: Post-transplant Ruxolitinib — Ruxolitinib will be given at a dose of 5 mg/kg twice daily starting at Day 30 post HCT, provided both the absolute neutrophil count (ANC) is > 1000/μl and platelet count is >30,000/μl.
  Arms: ACCEL-002
Drug: Supportive Care: Growth Factors — Granulocyte colony-stimulating factor (G-CSF) to accelerate neutrophil recovery should be administered starting at Day +5 with dose, route of administration, formulation, and duration of administration following institutional guidelines. Filgrastim biosimilars are permissible, but granulocyte-macrophage colony-stimulating factors are not permissible.
Procedure: Supportive Care: Blood Products — Transfusion thresholds for blood product support will be consistent with standard institutional guidelines. All blood products must be irradiated.
Other: Supportive Care: Infection Prophylaxis — Subjects should receive infection prophylaxis according to institutional guidelines and in accordance with the Center for Disease Control (CDC) guidelines49. Infection prophylaxis will include, but is not limited to, agents or strategies (e.g., polymerase chain reaction [PCR] screening and preemptive therapy) to reduce the risk of bacterial, viral (e.g., adenovirus, CMV, EBV, herpes simplex), opportunistic (e.g. Pneumocystis jirovecii, Toxoplasma gondii) and fungal (yeast and mold) infections.
  Infection risk should assess patient-, pathogen-, and immune-related factors that increase susceptibility to infection. Minimal parameters requiring prophylaxis include but are not limited to neutropenia (ANC≤500/μL), lymphopenia (ALC≤500/μL), and exposure to immunosuppression or GvHD. Use of intravenous immunoglobulin (IVIG) should be considered for total IgG<400 mg/dL during exposure to immunosuppression and/or GvHD.
Other: Supportive Care: Intravenous immune globulin (IVIG) — Intravenous immune globulin (IVIG) administration will be according to local institutional standard practice for hypogammaglobulinemia but is generally not recommended.
Drug: Supportive Care: Seizure prophylaxis — Subjects will receive busulfan seizure prophylaxis with levetiracetam, fosphenytoin, or lorazepam per institutional guidelines.
Other: Supportive Care: Monitoring and management of CRS — The use of HLA-mismatched PBSC has been associated with greater risk of CRS relative to bone marrow. Following the infusion of MMUD PBSC on Day 0, subjects should be monitored daily through Day 14 for the development of CRS. High index of suspicion is urged, particularly in the few days following infusion. Many sites have successfully intervened with tocilizumab in order to avoid severe or prolonged CRS. Supportive care is encouraged for CRS Grades 1-2 and tocilizumab (or alternative) is recommended for CRS grade 3-4 where subject outcome may be impacted (Appendix G - CRS Guidance and Management).
Other: Supportive Care: Prophylaxis against infections — Consider monitoring for EBV reactivation during abatacept treatment and continue for six months following HCT.
  Consider monitoring and prophylaxis for CMV infection/reactivation during abatacept treatment and for six months following HCT.
  Arms: ACCEL-001
Drug: Supportive Care: Prophylaxis against infections — For participants receiving ruxolitinib, the recommended maximum dose of fluconazole daily is 200 mg.
  Arms: ACCEL-002
Other: Supportive Care: Lipid elevations — Assess lipid levels 8-12 weeks from start of therapy with ruxolitinib and treat as needed.
  Arms: ACCEL-002
Other: Study treatment compliance — The administration of study agents must be recorded in the subject's medical chart for verification of study treatment compliance.
Other: Prohibited Concomitant Therapy — Prophylactic anti-viral cellular therapies and/or co-enrollment on studies using therapies for the prevention of GVHD is prohibited.
  Subjects reported to have received prohibited therapy while on this study will be withdrawn and will not be included in the primary and secondary analyses.
  No concomitant systemic immunosuppressive agents can be administered during PTCy (Day 3 and Day 4). If needed, administer at least 24 hours after completion of Day 4 PTCy.
  It is crucial that no systemic immunosuppressive agents are given until at least 24 hours after completion of the Day +4 dose of PTCy. This includes corticosteroids as anti-emetics but excludes tacrolimus and MMF. Steroid use is permitted as pre-medication prior to start of conditioning but is prohibited from Day 0 through 24 hours post Day 4 PTCy administration.
  If prohibited therapies are administered, these data must be reported in the study EDC on the Concomitant Medications form.
Other: Permitted Concomitant Therapy — Pre-medication and/or treatment for possible AEs related to PTCy are permitted. Subjects may continue all medications in compliance with local treatment center and local institutional guidelines, except those described in Section 7.9.1. If GVHD or infection occurs, enrollment on a clinical trial to treat infection or GVHD is permissible. At time of relapse, patients are permitted to enroll on a clinical trial or receive disease targeted therapy.
  The following medications/therapies must be reported on the study EDC Concomitant Medications form:
  * Medications taken to treat adverse events that have been reported on the study EDC Adverse Event form.
  * Antimicrobial prophylaxis (viral, bacterial, fungal, parasitic).
  * Antimicrobial pharmaceutical and cellular therapies used to treat grade II-III infections per BMT CTN grading criteria (Appendix D - BMT CTN Infection Grading).
  * Post HCT, primary malignant disease-directed pharmaceutical and cellular therapies.
  * Planned maintenance therapy
Other: Prohibited Concomitant Therapy — Treatment with any other Investigational Medicinal Product (IMP) is not allowed while on study treatment. An IMP is defined as any medication without any known FDA-approved indications.
  No other investigational drugs for GVHD are allowed.
  Arms: ACCEL-001
Other: Permitted Concomitant Therapy — Premedication and/or treatment for possible adverse events (AE)s related to abatacept are permitted.
  Arms: ACCEL-001
Other: Prohibited Concomitant Therapy — Treatment with any other Investigational Medicinal Product (IMP) is not allowed while on study treatment. An IMP is defined as any medication without any known FDA-approved indications.
  Concomitant use of ruxolitinib with fluconazole doses of greater than 200 mg daily should be avoided.
  No other investigational drugs for GVHD are allowed.
  Arms: ACCEL-002
Other: Permitted Concomitant Therapy — Premedication and/or treatment for possible AEs related to ruxolitinib are permitted.
  Arms: ACCEL-002

SUMMARY:
The purpose of this clinical trial is to compare drug combinations to learn which drugs work best to prevent graft-versus-host-disease (GVHD) in people who have received a stem cell transplant. The source of stem cells is from someone who is not related and has a different blood cell type than the study participant. The researchers will compare the new drug combination to a standard drug combination. They will also learn about the safety of each drug combination.

Participants will:

* Receive the standard or new drug combination after transplant
* Visit the doctor's office for check-ups and tests after transplant that are routine for most transplant patients
* Take surveys about physical and emotional well-being
* Give blood and stool samples.

DETAILED DESCRIPTION:
This platform protocol will evaluate the safety and efficacy of post-transplant cyclophosphamide (PTCy) based graft-versus-host disease (GVHD) prophylaxis after mismatched unrelated donor (MMUD) hematopoietic cell transplant (HCT). Participants with malignant hematologic diseases eligible per inclusion criteria, receiving MMUD peripheral blood stem cells (PBSCs) after myeloablative conditioning (MAC) or reduced-intensity conditioning (RIC) will be eligible to be enrolled by participating transplant centers. The platform protocol will estimate endpoints and provide a comparator arm for investigational interventional arms (ISAs).

Two investigational ISAs are part of the platform protocol - ACCEL-001 and ACCEL-002. The ISAs describe the specific features of the intervention being studied and treatment of participants assigned to that intervention, the specific target population, sample size required based on comparison to the control arm, specific study objectives, statistical methods for evaluating the interventions, and other specific intervention-related information and assessments. Additional ISAs may be added or closed throughout the lifetime of the trial.

ELIGIBILITY:
Inclusion Criteria, MAC RECIPIENTS:

1. Age 18 to < 66 years (chemotherapy-based conditioning) or < 61 years (TBI-based conditioning) at the time of signing informed consent
2. Patient or legally authorized representative has the ability to provide informed consent according to the applicable regulatory and institutional requirements
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Planned MAC regimen (see Table 8 in Section 7.4 for allowed MAC regimens)
5. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age 16-35
6. Product planned for infusion is MMUD T-cell replete PBSC as allograft
7. HCT-CI < 5 (Appendix H - Hematopoietic Cell Transplant Comorbidity Index Scoring). The presence of prior malignancy will not be used to calculate HCT-CI for this trial, to allow for the inclusion of patients with secondary or therapy-related AML or MDS.
8. One of the following diagnoses:

   1. AML, ALL, or other acute leukemia in first remission or beyond with ≤ 5% marrow blasts and no circulating blasts or evidence of extramedullary disease. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients with MDS with no circulating blasts and with < 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% vs 5-10% blasts in MDS). Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
9. Cardiac function: Left ventricular ejection fraction ≥ 45% based on most recent echocardiogram or multi-gated acquisition scan (MUGA) results
10. Estimated creatinine clearance ≥ 45mL/min calculated by equation
11. Pulmonary function: diffusing capacity of the lungs for carbon monoxide (DLCO) corrected for hemoglobin ≥ 50% and forced expiratory volume in first second (FEV1) predicted ≥ 50% based on most recent PFT results
12. Liver function acceptable per local institutional guidelines
13. KPS of ≥ 70% (Appendix I - Performance Status)

Inclusion Criteria, RIC/NMA RECIPIENTS:

1. Age ≥ 18 years at the time of signing informed consent
2. Patient or legally authorized representative has the ability to provide informed consent according to the applicable regulatory and local institutional requirements
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Planned NMA/RIC regimen (see
5. Table 9 in Section 7.4 for allowed NMA/RIC regimens)
6. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age 16-35
7. Product planned for infusion is MMUD T-cell replete PBSC allograft
8. One of the following diagnoses:

   1. Patients with acute leukemia or chronic myeloid leukemia (CML) with no circulating blasts, no evidence of extramedullary disease, and with < 5% blasts in the bone marrow. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients with MDS with no circulating blasts and with < 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% vs 5-10% blasts in MDS.) Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   3. Patients with chronic lymphocytic leukemia (CLL) or other leukemias (including prolymphocytic leukemia) with chemosensitive disease at time of transplantation.
   4. Higher-risk chronic myelomonocytic leukemia (CMML) according to CMML-specific prognostic scoring system or high-risk MDS/myeloproliferative neoplasms (MPN) not otherwise specified are eligible, provided there is no evidence of high-grade bone marrow fibrosis or massive splenomegaly at the time of enrollment.
   5. Patients with lymphoma with chemosensitive disease at the time of transplantation.
   6. Patients with primary myelofibrosis or myelofibrosis secondary to essential thrombocythemia, polycythemia vera or MDS with grade 4 fibrosis.
9. Cardiac function: Left ventricular ejection fraction ≥ 40% based on most recent echocardiogram or MUGA results with no clinical evidence of heart failure
10. Estimated creatinine clearance ≥ 45mL/min calculated by equation
11. Pulmonary function: DLCO corrected for hemoglobin ≥ 50% and FEV1 predicted ≥ 50% based on most recent PFT results
12. Liver function acceptable per local institutional guidelines
13. KPS of ≥ 60% (Appendix I - Performance Status)

Exclusion Criteria:

1. Suitable HLA-matched related or 8/8 high-resolution matched unrelated donor available
2. Subject unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
3. Subjects with a prior allogeneic transplant
4. Subjects with an autologous transplant within the past 3 months
5. Subjects who are breastfeeding or pregnant
6. Uncontrolled bacterial, viral or fungal infection at the time of the transplant preparative regimen
7. Concurrent enrollment on a GVHD prevention clinical trial
8. Subjects who undergo desensitization to reduce anti-donor HLA antibody levels prior to transplant
9. Patients who are HIV-positive with persistently positive viral load. HIV-infected patients on effective anti-retroviral therapy (ART) with undetectable viral load within 6 months are eligible for this trial. Patients with well-controlled HIV are eligible provided resistance panels are negative, the patient is compliant with ART, and their disease remains well controlled.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Graft-versus-host disease-free, relapse-free survival (GRFS) | 1 year post-HCT
  To compare GRFS following transplantation of a PBSC product from a MMUD between standard-of-care PTCy-based GVHD prophylaxis (the control arm) and the combination of reduced-dose PTCy, ruxolitinib, tacrolimus, and MMF.
Graft-versus-host disease-free, relapse-free survival (GRFS) | 1 year post-HCT
  To compare GRFS following transplantation of a PBSC product from a MMUD between standard-of-care PTCy-based GVHD prophylaxis (the control arm) and the combination of reduced-dose PTCy, abatacept, and tacrolimus.

SECONDARY OUTCOMES:
Graft-versus-host disease-free survival (GFS) | 1 year post-HCT
  To assess GFS for each of the treatment arms
Infection-free survival (IFS) | 1 year post-HCT
  To assess IFS for each of the treatment arms
Overall survival (OS) | 1 year post-HCT
  To assess OS for each of the treatment arms
Progression-free survival (PFS) | 1 year post-HCT
  To assess PFS for each of the treatment arms
Non-relapse mortality (NRM) | 1 year post-HCT
  To assess NRM for each of the treatment arms
Cumulative incidence of relapse and disease progression | 1 year post-HCT
  To assess the cumulative incidence of relapse and disease progression for each of the treatment arms
Cumulative incidence of neutrophil engraftment | 1 year post-HCT
  To assess the cumulative incidence of neutrophil engraftment for each of the treatment arms
Cumulative incidence of platelet engraftment | 1 year post-HCT
  To assess the cumulative incidence of platelet engraftment for each of the treatment arms
Primary graft failure (PGS) and secondary graft failure (SGF) | 1 year post-HCT
  To assess PGF and SGF for each of the treatment arms
Incidence of ≥ grade 2 infections | 1 year post-HCT
  To assess the incidence of ≥ grade 2 infections for each of the treatment arms (BMT CTN grades II-III infection; Grades 1 ("mild", generally not reported), 2 ("moderate") and 3 ("severe/life threatening"))
Donor cell engraftment | 1 year post-HCT
  To assess donor cell engraftment for each of the treatment arms
Cumulative incidence of aGVHD | 1 year post-HCT
  To assess the cumulative incidence of aGVHD for each of the treatment arms
Cumulative incidence of cGVHD | 1 year post-HCT
  To assess the cumulative incidence of cGVHD for each of the treatment arms
Incidence of cytokine release syndrome (CRS) | 1 year post-HCT
  To assess the incidence of CRS for each of the treatment arms

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford, Palo Alto, California
  - MD Anderson, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided